CLINICAL TRIAL: NCT03295487
Title: The Value of Local Estrogen After TVT_O anti_incontinence Surgery in Postmenopausal Females.
Brief Title: ToT and Estrogen in Postmenopausal Females
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, sarah mohamed hassan, lecturer of obstetrics and gynecology, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Saramohamed7880
Record Dates: First submitted 2017-09-20; First posted 2017-09-28 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Stress Urinary Incontinence; Postmenopausal Disorder
Keywords: post menopausal stress incontinence; local estrogen
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Active Comparator): post menopausal female with genuine stress incontinence treated by TVT-O and local estrogen cream for 3 months after surgery
  Interventions: Procedure: TVT-O
- Group B (Active Comparator): post menopausal female with genuine stress incontinence treated by TVT-O only
  Interventions: Procedure: TVT-O

INTERVENTIONS:
Procedure: TVT-O — transobturator tape has been applied to all the patients in the study,and local estrogen vaginal cream is only applied to patients in group A
  Other Names: local vaginal estrogen cream

SUMMARY:
To compare the subjective and objective outcomes of TVT-O procedure alone versus the same procedure followed by the use of premarin vaginal cream for 3 months in postmenopausal female with genuine stress incontinence.

DETAILED DESCRIPTION:
a randomized controlled trial comparing the effect of using local estrogen cream after tot in postmenopausal female

ELIGIBILITY:
Inclusion Criteria:

-menopause patients included in group A should have: no history of breast cancer, ovarian cancer or uterine cancer No history of blood clots or thromboembolism No history of heart disease or stroke No history liver disease. Endometrial thickness less than 5mm Have a normal mammogram

Exclusion Criteria:

* presence of urge or mixed incontinence .

Ages: 49 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
outcome of the surgery | immediately after surgery
  clinical and urodynamic test improvment of the stress incontinence
outcome of the surgery | 3 months after surgery
  clinical and urodynamic test improvment of the stress incontinence

SECONDARY OUTCOMES:
nocturia , | immediatly after surgery
  symptom and sign from the patients
frequency, | immediatly after surgery
  symptom and sign from the patients
denovo urgency | immediatly after surgery
  symptom and sign from the patients
denovo urgency | 3 months after surgery
  symptom and sign from the patients
nocturia | 3 months after surgery
  symptom and sign from the patients
frequency | 3 months after surgery
  symptom and sign from the patients

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr El Ainiy Hospital, Cairo, Egypt